CLINICAL TRIAL: NCT04263103
Title: A Phase 4 Randomized, Single-blind Study to Evaluate the Multi-media Training（SJ-RS-WL2015）Software Rehabilitating Ability of Binocular Functions in Hospitalized Adolescent Patients With Intermittent Exotropia After Eye Surgery
Brief Title: A Training Software (SJ-RS-WL2015) Rehabilitating Intermittent Exotropia Binocular Functions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Guangzhou Shijing Medical Software (Industry)
Collaborators: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GuangzhouShijingMS2020ITE
Record Dates: First submitted 2020-02-06; First posted 2020-02-10 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2020-02

CONDITIONS: Intermittent Exotropia
Keywords: Intermittent Exotropia

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group with SJ-RS-WL2015 (Experimental): Item code: SJ-RS-WL2015, a visual training software program, 15 minutes of one section, twice a day, and for 1 year
  Interventions: Other: SJ-RS-WL2015 visual training program software
- control group (No Intervention): No special treatment, but observation

INTERVENTIONS:
Other: SJ-RS-WL2015 visual training program software — It is a software with perceptual learning methods for binocular functions
  Other Names: SJ-RS-WL2015 visual training program
  Arms: Experimental group with SJ-RS-WL2015

SUMMARY:
Evaluating the effect of SJ-RS-WL2015 visual training program in children with intermittent exotropia after eye surgery, including the improvement of simultaneous perception (I binocular function), fusion (II binocular function), stereopsis (III binocular function).

DETAILED DESCRIPTION:
All the patients are after eye surgery for intermittent exotropia. All the participants with 20/20 or better visual acuity.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Intermittent Exotropia
* Must be after eye surgery for Intermittent Exotropia
* Baseline Deviation Range: Esotropia<=5△ or Exotropia<15△ after Eye Surgery
* Visual Acuity: >=20/20

Exclusion Criteria:

* A-V patterns deviations
* Abnormal oblique or vertical rectus
* Nystagmus
* Ophthalmoplegia
* Anisometropia >2.5D
* With other eye surgery history
* Mental disorder
* Neural disease
* Tumor
* Heart disease
* Hypertension
* Epilepsy
* Severe systemic disease
* With vision therapy history within 4 weeks
* Implanted electronic device
* In other researches within 4 weeks

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 92 (Actual)
Dates: Start 2019-12-09 (Actual); Primary Completion 2020-10-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Stereopsis at 12 months | 12 months
  Measured with Synoptophore and Titmus stereo test, respectively
Change from Baseline Fusion at 12 months | 12 months
  Measured with Worth 4-dot test and Synoptophore, respectively
Change from Baseline Simultaneous Perception at 12 months | 12 months
  Measured with Bagolini striated lens, Worth 4-dot test, and Synoptophore, respectively
Change from Baseline Stereopsis at 6 months | 6 months
  Measured with Synoptophore and Titmus stereo test, respectively
Change from Baseline Fusion at 6 months | 6 months
  Measured with Worth 4-dot test and Synoptophore, respectively
Change from Baseline Simultaneous Perception at 6 months | 6 months
  Measured with Bagolini striated lens, Worth 4-dot test, and Synoptophore, respectively
Change from Baseline Stereopsis at 3 months | 3 months
  Measured with Synoptophore and Titmus stereo test, respectively
Change from Baseline Fusion at 3 months | 3 months
  Measured with Worth 4-dot test and Synoptophore, respectively
Change from Baseline Simultaneous Perception at 3 months | 3 months
  Measured with Bagolini striated lens, Worth 4-dot test, and Synoptophore, respectively
Change from Baseline Stereopsis at 2 months | 2 months
  Measured with Synoptophore and Titmus stereo test, respectively
Change from Baseline Fusion at 2 months | 2 months
  Measured with Worth 4-dot test and Synoptophore, respectively
Change from Baseline Simultaneous Perception at 2 months | 2 months
  Measured with Bagolini striated lens, Worth 4-dot test, and Synoptophore, respectively
Change from Baseline Stereopsis at 1 month | 1 month
  Measured with Synoptophore and Titmus stereo test, respectively
Change from Baseline Fusion at 1 month | 1 month
  Measured with Worth 4-dot test and Synoptophore, respectively
Change from Baseline Simultaneous Perception at 1 month | 1 month
  Measured with Bagolini striated lens, Worth 4-dot test, and Synoptophore,

SECONDARY OUTCOMES:
Visual Acuity | one year
  by LogMAR Visual Acuity Chart
Change from Baseline Deviation Degree at 1 year | 1 year
  by Prism Test
Change from Baseline Refractive Error at 1 year | 1 year
  by Phoropter

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Guangzhou Shijing Medical Software Co., Ltd., Guangzhou, Guangdong
  - Zhongshan Ophthalmic center, Sun Yat-sen University, Guanzhou, Guangdong

IPD SHARING:
Plan to Share IPD: No